CLINICAL TRIAL: NCT00894738
Title: Biomarkers of Cardiometabolic Risk in Children Treated With Antipsychotics: A Preliminary Study of Direct Measures
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 56790
Record Dates: First submitted 2009-05-04; First posted 2009-05-07 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Mental Disorders
Keywords: pediatric; mental illness; antipsychotic; cardiometabolic risk; Antipsychotic agents; Mental disorders diagnosed in childhood
MeSH Terms: conditions — Mental Disorders; Neurodevelopmental Disorders | interventions — Absorptiometry, Photon; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Some routine blood tests to assess glucose and lipid control and liver function, as well as an additional hepatitis screen if subjects have a history of hepatitis. Approximately 42 ml (3 tablespoons) of blood will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- antipsychotic treated: Children with psychiatric diagnoses who are currently treated with antipsychotic medications.
  Interventions: Procedure: Testing (MRS, US, DEXA, blood tests)
- healthy control: Age- and gender-matched children who do not have a psychiatric diagnosis, are not taking antipsychotic medications, and are otherwise healthy.
  Interventions: Procedure: Testing (MRS, US, DEXA, blood tests)

INTERVENTIONS:
Procedure: Testing (MRS, US, DEXA, blood tests) — Magnetic Resonance Spectroscopy (MRS) of the liver to determine hepatic triglyceride content; ultrasound (US) of the carotid artery to determine intima-media thickness; dual energy X-ray absorptiometry (DEXA) to determine body composition; fasting lipids, fasting insulin, C-reactive protein, liver enzymes and fibrinogen levels.

SUMMARY:
The proposed study aims to begin the multi-step process of establishing the reliability and validity of hepatic triglyceride content (HTGC) and carotid artery intima-media thickness (IMT) as biomarkers of cardiometablic risk in children treated for mental illness. The distribution of HTGC and carotid IMT-proximate indicators of cardiometabolic risk-across a range of dual-energy X-ray absorptiometry (DEXA)-measured adiposity in children treated with antipsychotic agents will be characterized in comparison to healthy, untreated, non-psychiatric controls, in order to estimate effect sizes for future studies incorporating these markers. The ability of HTGC and IMT to predict cardiometabolic risk as measured by commonly-used laboratory tests, such as fasting lipids, liver function tests, C-reactive protein and serum fibrinogen, will be assessed.

DETAILED DESCRIPTION:
Carotid artery intima media wall thickness (IMT) is one of the most developed biomarkers of cardiometabolic risk, with established reliability and predictive validity, and has been utilized as a surrogate endpoint for cardiovascular disease progression in FDA-reviewed registration studies. This technique has also been used in children and adolescents without psychiatric disorders, indicating that changes in IMT are positively correlated with metabolic syndrome criteria. Magnetic Resonance Spectroscopy (1H MRS) to quantify hepatic triglyceride content (HTGC) is a promising new marker of cardiometabolic risk, especially given the importance of nocturnal circulating free fatty acids in the development of insulin resistance leading to type 2 diabetes. Fatty liver, related in part to obesity, is the most common liver abnormality found in children ages 2-19, with one in ten children manifesting signs of macrovascular steatohepatitis. 1H MRS is a well-established methodology used to measure HTGC that correlates well with liver biopsy results. This technique has been studied in obese children without psychiatric disorders, and is widely considered to be the optimal noninvasive means by which to measure HTGC. Unfortunately, neither of these promising methods have been applied to the study of cardiometabolic risk in children with psychiatric disorders.

It is important to now study these biomarkers in psychiatric populations, where individuals are subject to treatments that can increase risk. Our group is experienced in the application of sophisticated, gold standard techniques for measuring cardiometabolic risk in psychiatric populations, and is-to our knowledge-the only group in the US using sensitive methodologies like stable isotopomer euglycemic clamps to study the pathophysiology leading to diabetes and cardiovascular disease in the mentally ill. An important goal of studying these biomarkers is to ultimately determine which of the more commonly available conventional risk measures (e.g., lipid profiles, adiposity measures) can be used alone or in combination to accurately identify children at highest risk, to aid in the development and targeting of effective interventions.

ELIGIBILITY:
The inclusion criteria for the treatment group participants are: i) aged approximately 6-18 years; ii) BMI percentile between approximately 25 and 99; iii) otherwise healthy and meets DSM-IV criteria for one or more childhood onset psychiatric disorder, any type (determined by semi-structured Missouri Assessment of Genetics Interview for Children or MAGIC-described below and at the discretion of the PI), treated with an antipsychotic > approximately 12 weeks; iv) able to give assent and have a guardian that can provide informed consent; and v) no antipsychotic medication dose changes for approximately 1 month, and no other medication changes for 1 month prior to study enrollment.

The inclusion criteria for healthy controls are: i) aged 6-18 years; ii) BMI percentile between approximately 25 and 99 iii) otherwise healthy and at the PI's discretion do not meet DSM-IV criteria for any Axis I psychiatric illness; iv) not currently taking any medications; and v) able to give assent, and have a guardian that can provide informed consent.

The exclusion criteria are: i) active suicidality or a primary diagnosis of major depressive disorder; ii) any lifetime use of antipsychotics; individual subjects with a remote, brief prior antipsychotic exposure may be considered for enrollment on a case by case basis by the PI; iii) the presence of any serious medical disorder that may confound the assessment of relevant biologic measures or diagnoses, including: significant organ system dysfunction; endocrine disease, including type 1 or type 2 diabetes mellitus; coagulopathy; anemia; or acute infection; all based on PI discretion; iv) subjects regularly taking within the last 3 months any glucose lowering agent, lipid lowering agent, exogenous testosterone, recombinant human growth hormone, or any other endocrine agent that might confound substrate metabolism, oral glucocorticoids (glucocorticoid nasal spray and inhalers are permitted), sedating antihistamines (non-sedating antihistamines such as but not limited to Claritin (loratadine) and Zyrtec (cetirizine) are permitted), and certain mood stabilizing agents, as some medications may themselves worsen or otherwise alter weight gain, glucose and lipid regulation or otherwise make it difficult to assess the effects of the antipsychotic alone; (note that exposure to many psychotropic agents including stimulants and SSRI's is permitted in order to maintain the generalizability of the sample); v) IQ < 70 (based on school records and/or evaluation by clinician); vi) current substance abuse; vii) past history of, or current dyskinesia; viii) stimulant dosage significantly higher (per PI judgment) than the equivalent of approximately 2 mg/kg/day methylphenidate equivalent dose.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children ages 6-18 who are currently being treated for a psychiatric condition with an antipsychotic medication, and age- and gender-matched healthy controls who are not treated with an antipsychotic medication.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ginger E Nicol, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Antipsychotic-Treated: Children with psychiatric diagnoses who are currently treated with antipsychotic medications.
Period: Overall Study
Arm/Group | Antipsychotic-Treated | Healthy Control
Started | 25 | 19
Completed | 25 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antipsychotic-Treated | Healthy Control | Total
Number analyzed (Participants) | 25 | 19 | 44
Age, Continuous [Mean (Standard Deviation); unit: years]
  Pre-pubertal status, ages 6-11 | 10.3 (1.5) | 9.5 (1.6) | 9.9 (1.6)
  Post-pubertal status, age 12-19 | 14.7 (1.7) | 15.3 (1.0) | 15.0 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 19 | 15 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 13 | 22
  Not White | 16 | 6 | 22
Body Mass Index (BMI) Percentile [Mean (Standard Deviation); unit: Percentile] | 67.5 (28.4) | 58.9 (30.2) | 63.8 (29.2)
Blood Pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic | 111 (9) | 112 (13) | 111 (11)
  Diastolic | 69 (6) | 67 (8) | 68 (7)
Dual Energy X-ray Absorptiometry (DEXA) Total Percent Fat [Mean (Standard Deviation); unit: percent of total body fat] | 26.3 (11.1) | 24.1 (11.4) | 25.3 (11.2)
Carotid Intima Media Thickness (CIMT) [Mean (Standard Deviation); unit: mm] — Population: 1 participant is missing a CIMT.
  mm
    number analyzed (Participants) | 24 | 19 | 43
    (all) | 0.51 (0.05) | 0.52 (0.05) | 0.51 (0.05)
Intrahepatic Triglyceride Content (IHTG) [Mean (Standard Deviation); unit: percent of liver fat] — Population: 1 participant is missing a IHTG.
  percent of liver fat
    number analyzed (Participants) | 24 | 19 | 43
    (all) | 2.5 (3.0) | 1.6 (1.4) | 2.1 (2.5)
Vitamin D Level [Mean (Standard Deviation); unit: ng/mL] | 18.4 (5.4) | 22.1 (7.1) | 20.0 (6.4)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] | 88.0 (8.1) | 87.2 (7.3) | 87.7 (7.7)
Fasting Insulin [Mean (Standard Deviation); unit: uIU/mL] | 15.5 (16.8) | 11.0 (5.8) | 13.5 (13.3)
Fasting Lipids [Mean (Standard Deviation); unit: mg/dL]
  Total Cholesterol | 164.2 (24.9) | 149.7 (25.5) | 158.0 (25.9)
  High Density Lipoprotein (HDL) Cholesterol | 57.1 (12.7) | 54.1 (15.2) | 55.8 (13.7)
  Triglycerides | 68.6 (40.7) | 68.8 (24.7) | 68.7 (34.3)
  Low Density Lipoprotein (LDL) Cholesterol | 93.4 (19.1) | 81.7 (20.1) | 88.3 (20.1)
High Sensitivity C-Reactive Protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] — Population: 1 participant is missing a hs-CRP.
  mg/L
    number analyzed (Participants) | 24 | 19 | 43
    (all) | 1.52 (3.20) | 0.77 (1.02) | 1.19 (2.49)
Total Protein [Mean (Standard Deviation); unit: g/dL] | 7.4 (0.5) | 7.1 (0.5) | 7.2 (0.5)
Albumin [Mean (Standard Deviation); unit: g/dL] | 4.4 (0.3) | 4.4 (0.2) | 4.4 (0.3)
Alkaline Phosphatase [Mean (Standard Deviation); unit: IU/L] — Population: 1 participant is missing a Alkaline Phosphatase measure.
  IU/L
    number analyzed (Participants) | 24 | 19 | 43
    (all) | 220.3 (67.8) | 234.1 (106.5) | 226.3 (86.2)
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: IU/L] — Population: 1 participant is missing an ALT.
  IU/L
    number analyzed (Participants) | 24 | 19 | 43
    (all) | 20.5 (7.1) | 18.9 (6.6) | 19.8 (6.8)
Aspartate Aminotransferase (AST) [Mean (Standard Deviation); unit: IU/L] — Population: 1 participant is missing an AST value.
  IU/L
    number analyzed (Participants) | 24 | 19 | 43
    (all) | 29.0 (6.0) | 31.4 (10.5) | 30.0 (8.3)
Total Bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.35 (0.16) | 0.50 (0.52) | 0.41 (0.37)
Fibrinogen [Mean (Standard Deviation); unit: mg/dL] — Population: 1 participant is missing a Fibrinogen.
  mg/dL
    number analyzed (Participants) | 25 | 18 | 43
    (all) | 301.3 (72.7) | 269.0 (45.0) | 287.8 (64.0)

OUTCOME MEASURES:

1. Primary Outcome: Carotid Artery Intima-media Thickness Measured by Ultrasonography.
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Antipsychotic-Treated | Healthy Control
Number analyzed (Participants) | 24 | 19
millimeters | 0.508 (0.053) | 0.519 (0.048)
Statistical Analysis 1: Comparison: Antipsychotic-Treated vs Healthy Control; The null hypothesis is that mean DEXA total percent fat is similar between the two groups of interest. The primary statistical model consisted of treatment group as a 2-level factor (AP-Treated Vs Non-AP Treated) and DEXA total percent fat as a covariate. Carotid intima-media thickness (CIMT) was the dependent variable; Test type: Superiority or Other; p = 0.49, ANCOVA — The p-value listed is for DEXA total percent fat and is not adjusted for multiple comparisons. The alpha level was set to 5%

2. Primary Outcome: Intrahepatic Triglyceride Content (IHTG) Measure by Liver Magnetic Resonance Spectroscopy.
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Antipsychotic-Treated | Healthy Control
Number analyzed (Participants) | 24 | 19
percent | 2.48 (3.03) | 1.57 (1.37)
Statistical Analysis 1: Comparison: Antipsychotic-Treated vs Healthy Control; The statistical analysis consisted of treatment group as a 2-level factor variable and DEXA total percent fat as a covariate. An interaction term between treatment group and DEXA total percent fat was also generated. Hepatic triglyceride content was the dependent variable. DEXA total percent fat was found to be significant while treatment group and the interaction between treatment group and DEXA total percent fat were not significant; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: No adverse event data was collected since this was a cross-sectional study.
Arm/Group | Antipsychotic-Treated | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No